CLINICAL TRIAL: NCT04104737
Title: Spire Medical Health Tag Respiratory Rate Validation in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spire, Inc. (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR 2019-330
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Spire Medical Health Tag (Experimental): Spire Medical Health Tag is worn by all subjects The study is open label
  Interventions: Device: Spire Medical Health Tag

INTERVENTIONS:
Device: Spire Medical Health Tag — Collect data to validate the respiratory rate performance of the Medical Health Tag developed by Spire Health. The Medical Health Tag respiratory rate will be evaluated during non-motion conditions over the range a range of 5-50 breaths per minute via Reference EtCO2.
  A FDA cleared, GE Healthcare S5 Multi-parameter monitoring system with End Tidal Carbon Dioxide (EtCO2) and 3- lead ECG will be used for the Respiratory and Pulse Rate References.
  Other Names: GE Healthcare S5 Multi-parameter monitoring system; End Tidal Carbon Dioxide (EtCO2); 3- lead ECG

SUMMARY:
The primary purpose of this study is to conduct a Respiratory Rate accuracy validation comparing the Spire Medical Health Tag to a FDA cleared End Tidal Carbon Dioxide monitor Reference Standard (GE Datex-Ohmeda).

After IRB approval, a minimum of 20 healthy volunteer test subjects, 18 or older will be entered into this study designed to validate the accuracy of the respiratory rate feature of the Spire Medical Health Tag (Device Under Test).

The subjects will be selected to represent a range of body types including small, average, muscular, and large with a range of BMIs. Each subject will be connected to a FDA cleared EtCO2 monitor (GE Datex-Ohmeda) and will be instrumented with a mouthpiece or open system mask that allows for measurement of EtCO2 derived respiratory rate. A range of stable respiratory rates will be elicited from each volunteer test subject with the use of a paced breathing application on a mobile phone. Subjects will also be connected to a 3-lead ECG (GE Datex-Ohmeda) for the purpose of monitoring heart rate and comparing to the pulse rate measurements recorded by the Spire Medical Health Tag.

The respiratory rate and pulse rate will be measured simultaneously for the Reference and the Device Under Test.

DETAILED DESCRIPTION:
The purpose of this study is to collect data to validate the respiratory rate performance of the Medical Health Tag developed by Spire Health. The Medical Health Tag respiratory rate will be evaluated during non-motion conditions over the range a range of 5-50 breaths per minute via Reference EtCO2. A FDA cleared, GE Healthcare S5 Multi-parameter monitoring system with End Tidal Carbon Dioxide (EtCO2) and 3-lead ECG will be used for the Respiratory and Pulse Rate References. There are no risks or adverse device effects to be assessed. There are no contraindications for use in the proposed study / study population.

This study will focus on the respiratory rate, RR parameter. The Spire Medical Health Tag is investigational and has not been cleared by the FDA. The intended purpose of the device under test is spot-checking, non-invasive monitoring / logging of respiratory rate on humans. For this evaluation, the device will be run in a continuous data collection mode.

The study population will include 20 healthy competent adults, ages 18 years and older. The subject selection will be a mix of males and females with small to large physiques. The subjects must understand the study and consent to participate by signing the Informed Consent Form. The subjects must be healthy showing no evidence of medical problems as indicated by satisfactorily completing the health assessment form and passing the health screening. Eligible subjects need to meet all of the inclusion criteria and none of the exclusion criteria for participation.

It is expected that the data collection will take approximately 4-7 days to complete. There is no additional followup required for the investigation.

The data from the Device Under Test will be collected on an application installed on the iOS or Android mobile device separate from the reference equipment.

Multi-parameter monitor used during the study to observe a subject's vital signs include ECG tracing, heart rate, respiratory rate, and EtCO2 with capnograph.

* GE Healthcare S5 Compact Monitor, M-NESTPR module with ECG, and/or Multi-parameter monitor
* Portable oxygen tank, mask and ambu bag
* GE Healthcare (Datex-Ohmeda) 3900 TruTrak+ / OxyTip+ Oxy-F-UN or Oxy-AF Sensor and Oxy-OL3 cable (SpO2 monitoring)
* Blood pressure cuff and stethoscope

Currently the FDA defines respiration rate devices as Class II devices. The Device Under Test in this study is considered non-significant risk device.

There are no risks or adverse device effects to be assessed. There are no contraindications for use in the proposed study / study population.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent
* Subject is adult over 18 years of age
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker
* Male or female of any race

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Subjects with known respiratory conditions such as:

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * respiratory or lung surgery,
  * emphysema, COPD, lung disease
* Subjects with self-reported heart or cardiovascular conditions such as:

  * have had cardiovascular surgery
  * Chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
* Self-reported health conditions as identified in the Health Assessment Form

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent head injury within the last 2 months,
  * Cancer / chemotherapy
* Other known health condition, should be considered upon disclosure in health assessment form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
measurement of respiratory rate to the Reference | 60 seconds
  The endpoint of interest is accuracy as measured by the Accuracy root-mean-square (Arms) difference between the Device Under Test (DUT) and the Reference EtCO2 (Ref) for all stable respiratory periods

CONTACTS AND LOCATIONS:
Overall Officials: Dena Raley, BS, Study Director — CTO Clinimark LLC.
Locations (2):
- United States (2):
  - Spire, Inc., San Francisco, California
  - Arthur Cabrera, MD., Louisville, Colorado

IPD SHARING:
Plan to Share IPD: No
No plan to share individual data